CLINICAL TRIAL: NCT05164991
Title: Visuo-Tactile Integration and Body Ownership in the Human Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other); Eye Hospital Jules Gonin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-0111
Record Dates: First submitted 2021-10-29; First posted 2021-12-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Behavior and Behavior Mechanisms; Body Representation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR imaging (Experimental): The experiment is aimed to induce a virtual rubber hand illusion, in which the individuals can potentially experience an embodiment illusion
  Interventions: Behavioral: Visuo-tactile stimulations of the right hand

INTERVENTIONS:
Behavioral: Visuo-tactile stimulations of the right hand — Participants lay down in the magnetic resonance (MR) scanner are presented with visual stimuli (videos of the virtual rubber hand - visual stroking) simultaneously in real time with tactile stimuli (robotic stroking of the participant's hand - tactile stroking). An MR-compatible robot systematically provides the tactile stroking on the participant's hand. MR-compatible goggles show the visual stroking. Patterns of long and short robotic movements will be provided.

SUMMARY:
The present project exploits brain imaging and neuroscience robotics to investigate the role of quantifiable visual input on the relationship between visuo-tactile integration and body ownership (the feeling that "this" body belongs to "me").

DETAILED DESCRIPTION:
Observational study, fundamental research, multicentric, national. The analysis of questionnaires, self-reports, and brain imaging associated with the RHI is used to understand the influence of visual input on body ownership. To this aim, participants lay down in the magnetic resonance (MR) scanner (Figure 1B), are presented with visual stimuli (videos of the virtual rubber hand - visual stroking) simultaneously in real time with tactile stimuli (robotic stroking of the participant's hand - tactile stroking), and in combination or not with the measurement of autonomic arousal (GSR) associated with the observation of a video showing the virtual rubber hand in a threatening situation (e.g. a knife approaching the virtual hand - unconscious RHI effects). By means of structured questionnaires and semi-structured self-reports, participants (i) evaluate eventual sensations felt during the visuo-tactile stimulation and (ii) report the personal feelings and impressions about body ownership for the virtual rubber hand (conscious RHI effects).

ELIGIBILITY:
Inclusion Criteria:

* general health
* personal interest
* age between 18 and 55 years old
* fulfil standard guidelines for fMRI studies

Exclusion Criteria:

* history of seizures, epilepsy
* specific medications or treatment
* concomitant diseases (e.g. cardiopathy)
* pregnancy
* unexplained loss of consciousness
* chronic headaches
* neurological illnesses
* head concussion,
* presence of metal in the neck or head
* implanted medical devices
* drug abuse
* inability to give consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Neuro-behavioral changes associated with vision-dependent alterations of body ownership, measured via brain activity (fMRI) | Through study completion, an average of 2 years
  Analysis of objective measures of the RHI

SECONDARY OUTCOMES:
Subjective Experience via VAS scale | Through study completion, an average of 2 years
  To understand the variations of the body ownership, Visual Analogic Scale, values 0 to 7, 0 = no illusory body ownership, 7 = strong illusory body ownership
Automatic response (skin conductance) | Through study completion, an average of 2 years
  Measure of the skin conductance response (SCR, measured in siemens) during experiment runs, which is an indirect measure of sympathetic activity.
  Compare the blocks in which a pre-recorded visual threat (a video in which a hand is being pricked by a syringe needle) with baseline blocks and expect a higher SCR signal during "visual threat" blocks compared to the baseline. The SCR will be measured through a device connected to a dedicated laptop and electrodes that will be attached to the left index and middle fingers from participants. The SCR will be saved in log files and estimated a posteriori for each block using a general linear model and the weight regressors will be compared. There are no risks to the participants (since it is a passive measurement) the electrodes are compatible to the magnetic resonance environment.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Ionta, Professor, Principal Investigator — Fondation Asile des Aveugles, 1002, Lausanne
Locations (1):
- ETH Zurich, Rehabilitation Engeineering Laboratory, Zurich, Switzerland